CLINICAL TRIAL: NCT02595216
Title: Clinical Study to Evaluate the Performance of Profound System With Nominal Angle of 75° to the Skin's Surface for Submental Laxity
Brief Title: Treatment With the Profound System for Submental Laxity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Syneron Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DHF20161
Record Dates: First submitted 2015-10-29; First posted 2015-11-03 (Estimated); Last update posted 2017-04-06 (Actual); Status verified 2017-04

CONDITIONS: Submental Laxity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- all subjects (Experimental): All subjects in this study will receive a single Profound system treatment to the submental area with the profound device; subjects will return to four follow- up visits: 1 week post treatment, 1, 3 and 6 months post treatment.
  Prior to treatment, tissue will be treated with injected tumescence or local dermal infiltration solution according to the protocol.
  Interventions: Device: Profound System

INTERVENTIONS:
Device: Profound System — The Profound system is indicated for use in dermatologic and general surgical procedures for electrocoagulation and hemostasis, and the percutaneous treatment of submental laxity

SUMMARY:
Prospective clinical study to evaluate the Profound efficiency Up to 60 healthy adult volunteers, male or females, 18 to 70 years old. All subjects in this study will receive a single treatment to the submental area with the profound device; subjects will return to four follow- up visits: 1 week post treatment, 1, 3 and 6 months post treatment.

Prior to treatment, tissue will be treated with injected tumescence or local dermal infiltration solution according to the protocol.

DETAILED DESCRIPTION:
This study is a Prospective clinical study to evaluate the Profound device for submental laxity.

Up to a total of 60 healthy candidates, seeking treatment for submental laxity. Subjects will receive one Profound treatment targeted to both dermal and subcutaneous layer of the skin.

Before treatment (15-20 minutes) the tissue to be treated will be injected with tumescence solution.

Each subject will be followed for additional four (4) post treatment visits

ELIGIBILITY:
Inclusion Criteria:

1. Subjects seeking laxity treatment for submental area
2. Healthy female or male subjects ages 18 to 70 years of age
3. Informed consent process completed and signed consent
4. Willing to receive the proposed Profound treatment and follow the protocol
5. For female subjects: not pregnant or lactating;
6. either post-menopausal, surgically sterilized, or using a medically acceptable form of birth control at least 3 months prior to enrollment (i.e., oral contraceptives, contraceptive implant, barrier methods with spermicide or abstinence)
7. Willing to have photographs taken of the treated areas to be used de-identified in evaluations, publications and presentations

Exclusion Criteria:

1. Surgery or any other procedure for laxity in the last 6 months
2. Pregnant or planning to become pregnant, having given birth less than 3 months ago, and/or breast feeding
3. Known allergy to lidocaine or epinephrine or antibiotics
4. Active malignancy or history of malignancy in the past 5 years
5. Having any active electrical implant anywhere in the body, such as a pacemaker or an internal defibrillator
6. Suffering from significant concurrent illness, such as cardiac disorders, diabetes (type I or II), lupus, porphyria, or pertinent neurological disorders (i.e. any disease state that in the opinion of the Physician would interfere with the anesthesia, treatment, or healing process)
7. Having a known anticoagulative or thromboembolic condition or taking anticoagulation medications one week prior to and during the treatment course (to allow inclusion, temporary cessation of use as per the subject's physician discretion)
8. History of immunosuppression/immune deficiency disorders (including HIV infection or AIDS) or currently using immunosuppressive medications
9. Suffering from hormonal imbalance, whether related to thyroid, pituitary, or androgen
10. History of significant lymphatic drainage problems
11. History of cancer which required lymph node biopsy or dissection
12. Suffering from significant skin conditions in the treated areas or inflammatory skin conditions, including, but not limited to, open lacerations or abrasions, hidradenitis, or dermatitis of the treatment area prior to treatment (duration of resolution as per the Investigator's discretion) or during the treatment course
13. History of keloid scarring, abnormal wound healing and / or prone to bruising
14. History of epidermal or dermal disorders (particularly if involving collagen or microvascularity), including collagen vascular disease or vasculitic disorders
15. Use of isotretinoin (Accutane®) within 6 months of treatment or during the study
16. Systemic corticosteroid therapy 6 months prior to and throughout the course of the study
17. Dysplastic nevi in the area to be treated
18. Participation in a study of another device or drug within 3 month prior to enrollment or during this study, if treatments of wrinkles or laxity were involved
19. Subject has palpable lymphadenopathy at any visit. Standard palpation techniques will be used
20. Subjects with history of severe edema
21. As per the Investigator's discretion, any physical or mental condition which might make it unsafe for the subject to participate in this study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-09; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Evaluate the Performance of Profound system to the skin's surface for submental laxity | at 6 months
  using Fitzpatrick Wrinkle and Alexiades-Armenakas Laxity Scales

SECONDARY OUTCOMES:
safety of the profound single treatment by record of the Number, severity and type of adverse events | from day 0 until 6 months
  Number, severity and type of adverse events recorded
Investigator satisfaction | day 0, 1, 3, and 6 months
  assessed by Investigator
Subject Satisfaction | 1, 3, and 6 months
  by Subject questionnaire
Subject pain assessment | day 0 (treatment)
  using Numerical Scale Response (NSR)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Beaty, M.D., Principal Investigator — Beaty Facial Plastic Surgery
Locations (5):
- United States (5):
  - Premier Plastic Surgery, San Mateo, California
  - Gladstone Clinic, San Ramon, California
  - Mark Beaty, Alpharetta, Georgia
  - Coliseum Health System, Macon, Georgia
  - Dr. Richard Gentile, Boardman, Ohio

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ruiz-Esparza J. Nonablative radiofrequency for facial and neck rejuvenation. A faster, safer, and less painful procedure based on concentrating the heat in key areas: the ThermaLift concept. J Cosmet Dermatol. 2006 Mar;5(1):68-75. doi: 10.1111/j.1473-2165.2006.00226.x. PMID 17173575